CLINICAL TRIAL: NCT03984227
Title: Studying of New Signaling Pathway Targeting Systemic Lupus Erythematosus
Brief Title: New Signaling Pathway Targeting Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Ragab Mohamed Ibrahem, ASSISTANT LECTURER OF MEDICAL BIOCHEMISTRY, Assiut University
Other Study IDs: Systemic lupus erythematosus
Record Dates: First submitted 2019-05-28; First posted 2019-06-12 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-05

CONDITIONS: SLE

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Retained
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SLE patient group: SLE diagnosed patients between (18- 60) years old will be enrolled. All participants should met at least four of the American College of Rheumatology criteria (Hochberg, 1997). Disease activity will be assessed in accordance with the SLE Disease Activity Score (SLEDAI 2000 (SLEDAI-2K) (Ward et al., 2000).
  Interventions: Genetic: Taking peripheral blood samples
- control group: The control group will include age and sex matched healthy volunteers
  Interventions: Genetic: Taking peripheral blood samples

INTERVENTIONS:
Genetic: Taking peripheral blood samples — quantitative real-time polymerase chain reaction

SUMMARY:
Systemic lupus erythematosus is inflammatory autoimmune disease that affects over one million people in the United States. It has a higher prevalence and incidence rate among women compared with men, and among African Americans compared with Caucasians. Despite advances in treatment, standardized mortality rates in SLE remain three times higher than in the general population. The risk of mortality is significantly increased because of renal disease, cardiovascular disease, and infection.The etiology of SLE is multifactorial, with genetic predisposition, environmental factors and epigenetic alterations are involved. However, the molecular mechanisms underlying this systemic autoimmune response remain largely unknown. A key issue in the pathogenesis of lupus is how intracellular antigens become exposed and targeted by the immune system.

DETAILED DESCRIPTION:
Antinuclear antibodies play a direct role in pathogenesis by forming immune complexes. These complexes can either deposit in the kidney or stimulate cytokine production. Dead and dying cells can fill the blood with a plentiful supply of immune complex components in lupus. So cell death is a critical issue in the pathway to auto-reactivity. Pyroptosis is a new member of cell death list. It combines the release of pro-inflammatory mediators and nuclear molecules in a way that could drive lupus. Nod-like receptor pyrins-3, caspase-1, IL-18, and IL-1β are commonly accepted markers of pyroptosis.

Gasdermin D was recently identified as the final pyroptosis executioner downstream of inflammasome activation, and may be an attractive drug target for many diseases. GSDMD is a member of the gasdermin protein family. It was identified as a caspase substrate. Under normal cellular conditions, the C-terminus of GSDMD auto-inhibits the pore-forming activity of the N-terminus. When extracellular signals associated with pyroptosis activate inflammasomes they subsequently cleave and activate caspases-1, -4, -5, and -11. Consequently, activated caspase-1 cleaves and separates the N- and C-terminals of GSDMD. Activated GSDMD forms nanoscopic pores in the cell membrane, leading to the release of proinflammatory materials and cell swelling.

Reactive oxygen species regulates the signaling pathways in response to the changes of the intracellular and extracellular environments. However, overproduction of ROS is toxic and lead to dysfunction of cell and tissue. Oxidative stress is increased in SLE. The increased ROS could promote the release of inflammatory related signaling factors, including nod-like receptor inflammasome and nuclear factor-κB. A recent study showed that inhibition of ROS generation suppressed pyroptosis of hematopoietic stem cells. It has been widely reported that NF-kB is a critical molecular switch for cellular response to oxidative stress. NF-kB exists in the form of dimer and has been demonstrated to be involved in the development and progression of various diseases associated with inflammation, apoptosis, and proliferation. A recent study showed that NF-kB is an essential transcription factor of GSDMD.

In the recent decades, increasing evidence have revealed the roles of epigenetic dysregulation, including microRNA, in the pathogenesis of SLE. MiRNAs is a class of short non-coding RNA approximately 21-25 nucleotides in length that plays important roles in many cellular processes by regulating gene expression. MiRNAs make up a novel class of post-transcriptional gene regulators By combining with the 3' noncoding region of target gene mRNA inducing their degradation or impairing their translation.

MiR-379-5p is located at delta-like 1 homolog-deiodinase, iodothyronine 3 genomic region on 14q32.31. The DLK1-DIO3 region contains 54 miRNAs that is associated with organ development and disease pathogenesis, especially carcinogenesis. Luciferase reporter assays showed that GSDMD was a direct target of miR-379-5p. The over-expression of miR-379-5p blocked the arsenite induced increases of GSDMD levels effect that were reversed by up-regulation of GSDMD.

ELIGIBILITY:
Inclusion Criteria:

* SLE diagnosed patients between (18- 60) years old will be enrolled.

Exclusion Criteria:

* Patients with known pre-existing immunological disorders.
* Patients with known pre-existing infection.
* clinical diagnosis of cancer.
* patients diagnosed with concomitant acute myocardial infarction.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: - SLE diagnosed patients between (18- 60) years old will be enrolled. All participants should met at least four of the American College of Rheumatology criteria (Hochberg, 1997). Disease activity will be assessed in accordance with the SLE Disease Activity Score (SLEDAI 2000 (SLEDAI-2K) (Ward et al., 2000).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
determination of the expression levels of GSDMD, NF-kB and miR-379-5p in SLE group and Control group | 6 months
  GSDMD, NF-kB and miR-379-5p expression levels will be measured using quantitative real time PCR
detection of the relationship between oxidative stress and pyroptosis | 6 months
  correlation between oxidative stress and pyroptosis and detect if there is relationship between them

CONTACTS AND LOCATIONS:
Overall Officials: Ghada M Ezzat, PhD, Principal Investigator — Department of Medical Biochemistry, Faculty of Medicine, Assiut University; Marwa A Gaber, PhD, Principal Investigator — Department of Medical Biochemistry, Faculty of Medicine, Assiut University

REFERENCES:
- [Result] Basiorka AA, McGraw KL, Eksioglu EA, Chen X, Johnson J, Zhang L, Zhang Q, Irvine BA, Cluzeau T, Sallman DA, Padron E, Komrokji R, Sokol L, Coll RC, Robertson AA, Cooper MA, Cleveland JL, O'Neill LA, Wei S, List AF. The NLRP3 inflammasome functions as a driver of the myelodysplastic syndrome phenotype. Blood. 2016 Dec 22;128(25):2960-2975. doi: 10.1182/blood-2016-07-730556. Epub 2016 Oct 13. PMID 27737891
- [Result] Dang Y, Wang X, Hao Y, Zhang X, Zhao S, Ma J, Qin Y, Chen ZJ. MicroRNA-379-5p is associate with biochemical premature ovarian insufficiency through PARP1 and XRCC6. Cell Death Dis. 2018 Jan 24;9(2):106. doi: 10.1038/s41419-017-0163-8. PMID 29367615
- [Result] Li J, Xue J, Wang D, Dai X, Sun Q, Xiao T, Wu L, Xia H, Mostofa G, Chen X, Wei Y, Chen F, Quamruzzaman Q, Zhang A, Liu Q. Regulation of gasdermin D by miR-379-5p is involved in arsenite-induced activation of hepatic stellate cells and in fibrosis via secretion of IL-1beta from human hepatic cells. Metallomics. 2019 Feb 20;11(2):483-495. doi: 10.1039/c8mt00321a. PMID 30643918
- [Result] Magna M, Pisetsky DS. The Role of Cell Death in the Pathogenesis of SLE: Is Pyroptosis the Missing Link? Scand J Immunol. 2015 Sep;82(3):218-24. doi: 10.1111/sji.12335. PMID 26118732
- [Result] Shi G, Abbott KN, Wu W, Salter RD, Keyel PA. Dnase1L3 Regulates Inflammasome-Dependent Cytokine Secretion. Front Immunol. 2017 May 8;8:522. doi: 10.3389/fimmu.2017.00522. eCollection 2017. PMID 28533778